CLINICAL TRIAL: NCT03598530
Title: Fracture-Related Outcome Study for Operatively Treated Tibia Shaft Fractures (FROST)
Brief Title: Fracture-Related Outcome Study for Operatively Treated Tibia Shaft Fractures
Acronym: FROST
Status: Active, not recruiting | Type: Observational
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Collaborators: DePuy Synthes (Industry)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: FROST_RP_v3.0
Record Dates: First submitted 2018-07-12; First posted 2018-07-26 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Tibial Fracture; Fracture of the Tibia Type AO/OTA 42
Keywords: Fracture fixation; Surgical treatment; Fracture reduction
MeSH Terms: conditions — Tibial Fractures | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Tibial Shaft Fracture: Patients sustaining a tibial shaft fracture (AO/OTA type 42) that requires surgery
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Surgical fracture fixation, using osteosynthesis, including single or multiple staged procedures (e.g. primary External Fixation and later conversion to internal fixation).
  Other Names: Operative; Surgical treatment

SUMMARY:
Approximately 1000 patients presenting with tibial shaft fractures (AO type 42) will be enrolled prospectively in this registry. All patients are treated and followed at 6 weeks, 6 months and 1 year postoperative always following the local standard of care (routine) visit schedule up to 36 months if required.

Data collection includes patient and fracture details, treatment details, functional, clinical and patient-reported outcomes and anticipated or procedure- and implant-related adverse events (i.e. complications) and their corresponding treatment

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at the time of the injury
* Diagnosis of a primary tibial shaft fracture (fracture type 42 according to the AO/OTA Fracture and Dislocation Classification) that will be treated operatively as part of standard of care

Exclusion Criteria:

* Pathological fracture caused by malignancy
* Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years old that present a tibial shaft fracture (type 42 according to the AO/OTA Fracture and Dislocation Classification), resulting from a trauma and not caused by a malignancy, that requires surgical treatment.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient-reported outcome | 6 weeks / 6 months / 12 months / 36 months
  Change in PROMIS Pain interference (v1.0 - Pain Interference 8a) over the the follow-up period Change in PROMIS: Physical function (mobility) (v2.0 - Physical Function 10b) over the the follow-up period

OTHER OUTCOMES:
Time to bone healing/union | 6 weeks / 6 months / 12 months / 36 months
  Time elapsed between treatment and union evaluated clinically and radiologically.

CONTACTS AND LOCATIONS:
Overall Officials: Willem J Metsemakers, Prof., Principal Investigator — Department of Trauma Surgery, UZ Leuven
Locations (15):
- United States (3):
  - NYU Langone and affiliated Hospitals, New York, New York
  - NYU Langone Jamaica Hospital Medical Center, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Department of Trauma Surgery, UZ Leuven, Leuven, Belgium
- Germany (3):
  - University Medical Center Mainz, Mainz
  - Medical Faculty LMU Munich, Munich
  - University Hospital Münster, Münster
- Queen Mary Hospital, Hong Kong, Hong Kong
- Sengkang General Hospital, Singapore, Singapore
- Tygerberg Hospital, Cape Town, South Africa
- Korea University Guro Hospital, Seoul, South Korea
- Switzerland (2):
  - University Hospital Basel, Basel
  - University Hospital Zurich, Zurich
- United Kingdom (2):
  - University Hospitals Coventry & Warwickshire NHS Trust, Coventry
  - Leeds General Infirmary University Hospital, Leeds

IPD SHARING:
Plan to Share IPD: Undecided
Registry Steering Committee does accept request to access the data after a minimum of 200 patients have been enrolled and followed-up for at least 1 year.
  The Registry Steering Committee will share anonymized data. Charges may apply.

REFERENCES:
- [Derived] Metsemakers WJ, Kortram K, Ferreira N, Morgenstern M, Joeris A, Pape HC, Kammerlander C, Konda S, Oh JK, Giannoudis PV, Egol KA, Obremskey WT, Verhofstad MHJ, Raschke M; F.R.O.S.T. Study Group. Fracture-related outcome study for operatively treated tibia shaft fractures (F.R.O.S.T.): registry rationale and design. BMC Musculoskelet Disord. 2021 Jan 9;22(1):57. doi: 10.1186/s12891-020-03930-x. PMID 33422025